CLINICAL TRIAL: NCT03071042
Title: A Phase I Dose Escalation Clinical Trial of Apatinib Tablets Plus Docetaxel as Second-line Treatment in Locally Advanced or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: A Clinical Trial of Apatinib Plus Docetaxel in Locally Advanced or Metastatic Gastric or GEJ Adenocarcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hongming Pan, MD, Principal Investgator, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-G306
Record Dates: First submitted 2016-02-14; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-02

CONDITIONS: Metastatic Gastric Adenocarcinoma
MeSH Terms: interventions — apatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib plus Docetaxel (Experimental): Each subject will receive one dose of Apatinib in the whole cycle (21 days), during which single dose induced DLT and safety monitoring will be performed. If the initial dose is well tolerated, next cycle the subject will receive more Apatinib as respectively. This study will enroll in 4 cohorts of Apatinib; cohort 1 at the dose of 425mg Apatinib, which followed by cohort 2(500mg), cohort 3(675mg) and cohort 4(750mg).
  Interventions: Drug: Apatinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Apatinib — Apatinib Mesylate Tablets 425mg (500mg，675mg or 750mg) po. qd continuous;
  Other Names: YN968D1,(AiTan®)
Drug: Docetaxel — Docetaxel 60mg/m2 ivgtt day 1, q21d Combined use of Docetaxel and Apatinib
  Other Names: Aisu®

SUMMARY:
This study evaluated the tolerance, safety and efficacy of Apatinib plus Docetaxel as the second-line treatment in locally advanced or metastatic gastric cancer (including Gastroesophageal junction (GEJ) Adenocarcinoma).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has to voluntarily join the study and sign the Informed Consent Form for the study;
2. Age: ≥18 years old;
3. Locally advanced or metastatic gastric cancer (including Gastroesophageal junction (GEJ) Adenocarcinoma ) patients confirmed by radiologic imaging or endoscopy tests, who had failed in first-line treatments;

   * First-line treatment should be 5-Fu combined with platinum based regimen;
   * Adjuvant/neoadjuvant chemotherapy should be defined as the first-line treatment, if recurrence happened within 6 months after completion of 5-Fu and platinum based adjuvant/ neoadjuvant chemotherapy;
4. Adjuvant/neoadjuvant chemotherapy history is allowed, if first-line treatment is applied more than 6 months later than prior treatments;
5. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure;
6. ECOG Performance Status ≤1;
7. Life expectancy shouldn't less than 16 weeks, since the first medicine application time;
8. Major organ function has to meet the following criteria (within 28 days before treatment):

   * HB ≥9.0 g/dL
   * ANC ≥1.5X109/L
   * PLT ≥100x109/L
   * Bilirubin ≤1.5 times the upper limit of normal (ULN)
   * ALT (SGOT) and AST (SGPT) ≤2.5 × ULN, unless liver metastases; if any, the ALT and AST≤5 × ULN
   * Serum Cr ≤ 1.5 x ULN
9. Patients must have at least one assessable lesion (including measurable and/or immeasurable) by radiological imagine (CT/MRI);
10. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 28 days before enrollment and the test result must be negative. Or menopause women, defined as follow:

    * ≥1 year no menstruation, after abort exogenous hormone treatment
    * Serum LH and FSH meet menopause criteria
    * More than 1 year no menstruation for ovarian function failure induced by radiation therapy.
    * More than 1 year no menstruation for menopause induced by chemotherapy
    * Surgical sterilization accepted (hysterectomy or ovariectomy)

Exclusion Criteria:

1. Involved in another on-going clinical trials;
2. Accept more than one chemotherapy previously in advanced gastric cancer (except more than 6 months from adjuvant/neoadjuvant treatment);
3. Prior taxane treatment (including Paclitaxel and Docetaxel);
4. Prior VEGFR inhibitor treatment (including Sorafenib and Sunitinib);
5. History of another malignancy within the last five years except cured nonmelanoma Skin cancer and carcinoma in situ of uterine cervix;
6. Any factors that influence the usage of oral administration;
7. History of the investigational agent treatment in 14 day prior to enroll in study (longer time period may be required which depends on drug characteristic);
8. Accept any chemotherapy and radiotherapy (excluding Palliative radiotherapy) in 3 weeks prior to study (longer time period may be required which depends on drug characteristic);
9. Poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than Class I; I-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class I cardiac dysfunction; Patients with positive urinary protein;
10. Poor-controlled adverse events (excluding Alopecia) induced by tumor therapy (>class 1 CTCAE);
11. History of intestinal obstruction or more than class 3 or 4 (CTCAE) gastrointestinal bleeding in 4 weeks prior to enroll in study;
12. Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
13. Clinical evidence in central nervous system (CNS) and poor-controlled CNS metastasis (No necessary to confirm negative CNS metastasis by CT/MRI);
14. Surgery within 2 weeks prior to enroll in study;
15. History of significant and poor-controlled diseases or infection, in the opinion of investigators, may impact the safety of the patients of the study;
16. Known history of human immunodeficiency, e.g. HIV positive;
17. Known or suspected allergy to the investigational agent or any agent given in association with this trial;
18. Pregnant or lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Tolerance profile of participants with treatment-related adverse events as assessed by CTCAE v4.0 | At least 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hongming Pan, MD, Study Chair — The Affiliated Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided